CLINICAL TRIAL: NCT02953119
Title: Prehabilitation for Elective Major Abdominal Surgery: a Randomised Controlled Trial
Brief Title: Prehabilitation for Elective Major Abdominal Surgery
Acronym: PISO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Nicolas DEMARTINES (Other)
Responsible Party: Sponsor-Investigator, Nicolas DEMARTINES, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 469/15
Record Dates: First submitted 2016-10-18; First posted 2016-11-02 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): The patients will undergo an exercise test on a cycle ergometer (VO2 max), a grip strength test (Jamar dynamometer), a Time Up and Go (TUG) test and a 6 Minutes Walking Test (6-MWT), before and after prehabilitation. Intervention involves 3 training sessions per week during 3 weeks preoperatively, according to the high intensity interval training model, wich consists of:
  * 5 minute warm-up (50% of Cardiopulmonary exercise testing, CPET)
  * Two 10 minute series of 15 sec sprint intervals (100%) interspersed by 15 sec pauses and a 4 min rest between the two series
  * Cool down with a 5 min active recovery period (30%) The grip strength test (Jamar dynamometer), TUG-test and 6-MWT will be repeated between 4 and 6 weeks and 8 and 10 week postoperatively.
  Interventions: Other: Prehabilitation
- Controls (No Intervention): The patients will also undergo an exercise test on a cycle ergometer, a grip strength test (Jamar dynamometer), a TUG-test and a 6-MWT, but only once preoperatively, and between 4 and 6 weeks and 8 and 10 week postoperatively.

INTERVENTIONS:
Other: Prehabilitation
  Arms: Prehabilitation

SUMMARY:
Prehabilitation is a concept that challenges the traditional models of recovery by initiating the recovery process preoperatively. Improvement of physical capacity by means of prehabilitation may facilitate better recovery after surgery.

The aim of the present study is to evaluate the impact of preoperative physical exercise training (prehabilitation) on postoperative recovery and clinical outcomes after major abdominal surgery.

DETAILED DESCRIPTION:
Major abdominal surgery is a great stressor to patients and causes large physiological changes, leads to tissue trauma, immobility, psychological distress and reduced quality of life. Physical capacity appears to be an important predictor for postoperative recovery after major abdominal surgery. Prehabilitation is a concept that challenges the traditional models of recovery by initiating the recovery process preoperatively. Improvement of physical capacity by means of prehabilitation may facilitate better recovery after surgery. More specifically prior to major abdominal surgery, preoperative exercise therapy is associated with improved physical fitness of patients, but whether or not this results in fewer complications or faster convalescence remains unclear.

The aim of the present study is to evaluate the impact of preoperative physical exercise training (prehabilitation) on postoperative recovery and clinical outcomes after major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

Elective major abdominal surgery:

* Esophagus, stomach
* Liver, pancreas
* Small intestine, colon, rectum
* Benign or malignant disease
* Other intra-abdominal open or laparoscopic surgery lasting> 2 hours
* Delay of 3 weeks between consultation and surgery

Exclusion Criteria:

* Patient < 18 years, consent not obtained
* Coronary artery disease (≥ stage III according to CCS)
* Heart disease (≥ stage III according to NYHA)
* Uncontrolled cardiac arrhythmias
* COPD (GOLD stage ≥ III)
* Physical inability to ride a bike
* Orthopedic surgery in the last 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | Up to 30 postoperative days
  Comprehensive Complication Index (CCI)

SECONDARY OUTCOMES:
Postoperative most severe complication | Up to 30 postoperative days
  Clavien classification
Length of stay | Up to 30 postoperative days
  From the day of hospitalization to the exit
Readmission rates | Up to 30 postoperative days
  Any readmission to the hospital
Exercise capacity | At 3 and 1 week preoperatively
  Exercise testing on a cycloergometer(VO2 max)
Life satisfaction | At 3 and 1 week preoperatively, then at 4 and 8 weeks postoperatively
  Specific questionnaire (EORTC:European Organisation for Research and Treatment of Cancer)
Biological inflammatory response | Up to 3 postoperative days
  C-reactiv protein (CRP) measure
Exercise capacity | At 3 and 1 week preoperatively, then at 4 and 8 weeks postoperatively
  Time up and go test
Walking capacity | At 3 and 1 week preoperatively, then at 4 and 8 weeks postoperatively
  6 minutes Walking Test
Happiness | At 3 and 1 week preoperatively, then at 4 and 8 weeks postoperatively
  Specific questionnaire (EMMBEP questionnaire)
Nutritional response | Up to 3 postoperative days
  Albumin measure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hübner, Principal Investigator — University Hospital CHUV
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michel A, Gremeaux V, Muff G, Pache B, Geinoz S, Larcinese A, Benaim C, Kayser B, Demartines N, Hubner M, Martin D, Besson C. Short term high-intensity interval training in patients scheduled for major abdominal surgery increases aerobic fitness. BMC Sports Sci Med Rehabil. 2022 Apr 7;14(1):61. doi: 10.1186/s13102-022-00454-w. PMID 35392968